CLINICAL TRIAL: NCT06737809
Title: HIPrevision - A Randomized Multicenter Clinical Investigation of Antimicrobial IP-Coated Revision Hip Prostheses
Brief Title: IP-coated Revision Hip Implants
Acronym: HIPrevision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-G-H-2023; CIV-24-05-047447 (Other: EUDAMED)
Record Dates: First submitted 2024-11-19; First posted 2024-12-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Peri-Prosthetic Joint Infection
Keywords: arthroplasty; replacement; hip; anti-infective agent; silver; periprosthetic joint infection
MeSH Terms: interventions — Microscopy, Electron, Scanning Transmission; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IP coated hip arthroplasty implants (Experimental): Participants receive an infection prevention (IP) coated hip implant
  Interventions: Device: IP Plasmafit® Revision cup (and stem) system
- Standard hip arthroplasty implants (Active Comparator): Participants receive a standard (uncoated) hip implant
  Interventions: Device: IP Plasmafit® Revision cup (and stem) system

INTERVENTIONS:
Device: IP Plasmafit® Revision cup (and stem) system — Revision total hip arthroplasty (THA) due to periprosthetic joint infection

SUMMARY:
The primary aim of the clinical investigation is to demonstrate the efficacy of a silver-based antimicrobial coating on hip implants in the reduction of periprosthetic infections in revision hip arthroplasty due to periprosthetic infection.

DETAILED DESCRIPTION:
The clinical investigation will include patients indicated for revision hip arthroplasty due to chronic periprosthetic infection. Subjects will either receive standard CE-marked revision hip implants or the newly developed IP (Infection prevention)- coated revision hip implants. The primary clinical benefit of the IP hip implant components remains the functional restoration of the hip joint and pain relief, as successfully shown for the uncoated predecessor devices, but additionally the IP coating is regarded ancillary to the intended purpose of the implant. Periprosthetic infections are one of the major complications in revision hip arthroplasty, leading to implant re-revision. A clinical investigation to evaluate additional measures to reduce this complication rate in revision total hip arthroplasty therefore has high clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients indicated for unilateral cementless acetabular and hip stem revision due to chronic periprosthetic infection (according to EBJIS definition): single-stage or two-stage surgical procedure according to clinical standard at the clinical investigation site
* According to the assessment of the clinical investigator, the subject is therapy compliant and able to attend the follow-up visits
* ASA physical status I - III
* Patient's signed written informed consent is available

Exclusion Criteria:

* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)
* The investigational implant components (femoral and/or acetabular) are not suitable for the patient anatomy or bone defect
* Patients who require plate osteosynthesis at the implantation site
* Patients with an already implanted silver-coated device
* Patients with immunodeficiency, i.e. patients currently receiving immunosuppressive therapy or patients with severe immunodeficiency requiring drug therapy
* Patients currently undergoing cancer treatment, e.g. chemotherapy or radiation therapy
* Severe soft tissue defects that require local or free flap procedure
* Periprosthetic joint infections with evidence of fungal infection
* Antibiotic suppression therapy
* BMI > 40 kg/m2
* Pregnancy, breast-feeding, or women of childbearing potential and not taking adequate contraceptive precautions
* Known or patient reported hypersensitivity to silver or titanium
* Patients held in a custodial setting
* Patients in a relationship of dependence on the sponsor, the clinic or the investigator
* Patients with contraindication for the investigational and comparator devices:
* in case of secondary diseases influencing the function of the joint implant
* in case of severe osteoporosis or osteomalacia
* in case of poor bone quality and osseous malformations, diseases in the area of the implant fixation, which may primarily or subsequently affect the stability of the joint replacement anchorage
* in case of non-regenerative bone conditions with lack of proximal femoral bone support and failure of defect union when use of prosthesis heads with neck length XXL is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of periprosthetic joint infections | 12 months
  Participants are monitored for 12 months after revision surgery. Every case of periprosthetic joint infection according to the definition of the EBJIS classification counts.

SECONDARY OUTCOMES:
Change of functional outcome over follow-up period (Harris Hip Score (HHS)) | 2 years post operative
  Harris-Hip-Score: The Harris Hip Score (HHS) is a clinical tool used to evaluate the function of the hip joint, particularly after hip surgery or in cases of hip disease.
  The HHS consists of 10 items divided into four categories:
  Pain (maximum 44 points) Function (maximum 47 points) Range of Motion (maximum 5 points) Deformity (maximum 4 points)
Changes in quality of life | 2 years post operative
  Measure Description: EQ-5D-5L
  The EQ-5D-5L is a standardized instrument used to measure health outcomes. Developed by the EuroQol Group (EQ), it assesses five dimensions (5D) of health:
  Mobility Self-care Usual activities Pain/discomfort Anxiety/depression Each dimension has five levels (5L) of severity: no problems, slight problems, moderate problems, severe problems, and extreme problems
Implant survival | 2 years post operative
  Measure Description: Kaplan-Meier implant survival Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period. The revision-free survival rate is the performance indicator of the product under investigation and confirms the clinical outcome of the hip prosthesis. Information on survival of the implant will be collected until the last follow-up of the study patients took place.
Radiographic assessment | 2 years post operative
  radiographic measurements to assess implant migration, signs of loosening and changes in the fixation area over time
Occurrence of safety issues with the new device | 2 years post operative
  Adverse events, device failures and component revision will be monitored throughout the study to assess the safety
Level of silver ion concentration | 12 months
  Laboratory analysis will be performed to monitor silver ion concentration in biospecimen.
Changes in blood biomarkers for liver function | 12 months
  Participants will be monitored for their level of liver enzymes (ALT, AST, GGT)
Changes in blood biomarker for kidney function | 12 months
  Participants will be monitored for their level of kidney marker (eGFR).
Changes in blood biomarker for inflammation | 12 months
  Participants will be monitored for their level of inflammation marker CRP.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Meller, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Gruca Orthopedic and Trauma Teaching Hospital, Samodzielny Publiczny Szpital Kliniczny im. prof. Adama Grucy CMKP, Otwock, Poland